CLINICAL TRIAL: NCT04561479
Title: Evaluation of the Effects of Pulmonary Rehabilitation in Patients With Chronic Fibrotic Hypersensitivity Pneumonitis
Brief Title: Pulmonary Rehabilitation in Patients With Chronic Fibrotic Hypersensitivity Pneumonitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeliha ÇELİK, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 283
Record Dates: First submitted 2020-09-13; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Hypersensitivity Pneumonitis; Extrinsic Allergic Alveolitis
Keywords: Hypersensitivity Pneumonitis; Exercise Tolerance; Physical Activity; Muscle Strength
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Active Comparator): Intervention:Training group will receive upper extremity aerobic exercise training, inspiratory muscle training and progressive resistance training
  Interventions: Other: Pulmonary Rehabilitation
- Control Group (Sham Comparator): Control group will receive alternative upper extremity exercises and breathing exercises.
  Interventions: Other: Alternative Exercises

INTERVENTIONS:
Other: Pulmonary Rehabilitation — All exercise program will be applied during supervised session by a physiotherapist. Range of maximal heart rate will be screened by heart rate monitor during supervised session. Training group will receive upper extremity aerobic exercise training using arm ergometer at 60-80% of maximal heart rate (dyspnea perception at 3-4 level as well as fatigue perception at 5-6 level according to Modified Borg Scale). Inspiratory muscle training (Powerbreathe® Wellness-Inspiratory Muscle Trainer) at 50-60% of maximal inspiratory pressure (MIP) and progressive resistance training at 30-60% of 1 RM (using proprioceptive neuromuscular facilitation techniques (flexion, abduction, external rotation/extension, adduction, internal rotation) for upper extremity resistance training; using sandback for knee extensors) will be performed during 24 sessions (3 day/week; 8 weeks)
  Arms: Training Group
Other: Alternative Exercises — Control group will receive alternative upper extremity exercises combined with breathing exercises. Control group will perform alternative upper extremity exercises combined with breathing exercises during 3 days/week, for 8 weeks
  Arms: Control Group

SUMMARY:
The aim is to evaluate exercise capacity, respiratory functions, respiratory and peripheral muscle strength, inspiratory muscle endurance, physical activity level, quality of life, fatigue, dyspnea, anxiety, depression and investigate the impact of 24-session pulmonary rehabilitation training on these parameters in patients with chronic fibrotic hypersensitivity pneumonitis.

DETAILED DESCRIPTION:
Hypersensitivity pneumonitis is a syndrome that results in the excessive immune response to inhalation of various antigenic particles in the environment. Patients often experience irreversible physiological disorders and severe dyspnea in the future. Common disorders in these patients are lung function abnormalities, decreased exercise capacity, muscle weakness, oxygen diffusion limitation, impaired quality of life, physical inactivity and fatigue. The aim of this study is to evaluate the effects of pulmonary rehabilitation training on exercise capacity, dyspnea, respiratory functions, respiratory and peripheral muscle strength, inspiratory muscle endurance, physical activity level, quality of life, fatigue, dyspnea, anxiety, depression in patients with chronic fibrotic hypersensitivity pneumonitis. The study was planned as a prospective, double-blind, case-control study. At least 30 patients with hypersensitivity pneumonitis will be included in the study. The cardiopulmonary rehabilitation program will be included inspiratory muscle training, upper extremity aerobic exercise and progressive resistance training will be performed in the exercise training group during 24 sessions. Alternative upper extremity exercises combined with breathing exercises will be performed in the control group. Functional exercise capacity, respiratory functions, respiratory and peripheral muscle strength, inspiratory muscle endurance, physical activity levels, quality of life, fatigue, dyspnea, anxiety and depressions will be evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable
* Under standard medication
* 18-80 years of age
* Patients diagnosed with chronic fibrotic hypersensitivity pneumonitis

Exclusion Criteria:

* Having another diagnosed respiratory or cardiac problem
* Orthopedic, or neurological psychiatric diseases with a potential to affect functional capacity,
* Having a skeletal-muscular disease that may affect evaluation results
* Uncontrolled asthma, MI (myocardial infarction) in the last 4 weeks, unstable AP (angina pectoris), 2-3. degree block, rapid ventricular or atrial arrhythmias, ventricular aneurysm, acute systemic disorders (ARF (acute renal failure), thyrotoxicosis, infection), cooperation problem, severe aortic stenosis, dissecting aneurysm, uncontrolled CHF (chronic heart failure), uncontrolled hypertension ventricular aneurysm, severe pulmonary hypertension, thrombophlebitis / intracardiac thrombus, recent systemic/pulmonary embolism, acute pericarditis, endocarditis, myocarditis
* Cognitive disorders
* Patients who have contraindications for exercise testing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximal exercise capacity | Second day
  Maximal exercise capacity will be evaluated symptom limited cardiopulmonary exercise testing. The cardiopulmonary exercise test will be performed on the treadmill at a progressively increasing speed and grade.
Functional exercise capacity | First day
  Functional exercise capacity will be evaluated with 6-minute walking test according to the American Thoracic Society and European Respratory Society criteria
Oxygen consumption | Second day
  Oxygen consumption will be measured by cardiopulmonary exercise test.

SECONDARY OUTCOMES:
FEV1 | First day
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. FEV1 will be evaluated. The percentage of predicted value <70% will be expressed as abnormal
FVC | First day
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. FVC will be evaluated. The percentage of predicted value <70% will be expressed as abnormal
FEV1/FVC | First day
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. FEV1/FVC will be evaluated.
PEF | First day
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. PEF will be evaluated. The percentage of predicted value <70% will be expressed as abnormal
FEF2575 | First day
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respratory Society criteria. FEF2575 will be evaluated. The percentage of predicted value <50% will be expressed as abnormal
Respiratory muscle strength | First day
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device .
Inspiratory muscle endurance | First day
  It will be evaluated incremental threshold loading test, in which participants started an initial load of 30% of maximal inspiratory pressure with a 10% increment every 2 minutes.
Peripheral muscle strength-upper extremity | First day
  Upper extremity muscle strength will be evaluated using portable hand held dynamometer.
Peripheral muscle strength-lower extremity | First day
  Knee extensor muscle strength will be evaluated using portable hand held dynamometer.
Physical activity level | Three consecutive day
  Physical activity level will be evaluated multi sensor activity monitor for 3 consecutive days.
Disease Specific Quality of Life | Second day
  Quality of Life using St. George's Respiratory Questionnaire (SGRQ) will be evaluated. Scores range from 0 to 100, with higher scores indicating more limitations.
Fatigue | Second day
  Fatigue using Fatigue Severity Scale (Turkish version) will be evaluated. The scale comprises nine statements.The scale of possible responses are ranging from 1 (strongly disagree) to 7 (strongly agree). FSS total scores are usually reported as the mean score over the nine items; a higher score indicates greater severity.
Dyspnea during daily living activities | Second day
  Dyspnea using Modified Medical Research Council (MMRC) dyspnea scale will be evaluated. Modified Medical Research Council Dyspnea Scale, levels are graded as 0-4, higher scores imply higher dyspnea.
Anxiety | Second day
  Anxiety using Hospital Anxiety and Depression Scale will be evaluated. HADS consists of two subscales including anxiety and depression. Possible scores are ranged from 0 to 21 for each of the two subscales. The HADS manual indicates that a score between 0 and 7 is "normal," between 8 and 10 "mild," between 11 and 14 "moderate," and between 15 and 21 "severe."
Depression | Second day
  Depression using Hospital Anxiety and Depression Scale will be evaluated. HADS consists of two subscales including anxiety and depression. Possible scores are ranged from 0 to 21 for each of the two subscales. The HADS manual indicates that a score between 0 and 7 is "normal," between 8 and 10 "mild," between 11 and 14 "moderate," and between 15 and 21 "severe."

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha ÇELİK, MSc, Principal Investigator — Gazi University; Betül YOLERİ, PT, Principal Investigator — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof, Study Director — Gazi University; Haluk TÜRKTAŞ, Prof, Principal Investigator — Gazi University

REFERENCES:
- [Background] Dias OM, Baldi BG, Ferreira JG, Cardenas LZ, Pennati F, Salito C, Carvalho CRR, Aliverti A, Pereira de Albuquerque AL. Mechanisms of exercise limitation in patients with chronic hypersensitivity pneumonitis. ERJ Open Res. 2018 Aug 22;4(3):00043-2018. doi: 10.1183/23120541.00043-2018. eCollection 2018 Jul. PMID 30151370
- [Background] Dowman LM, McDonald CF, Hill CJ, Lee AL, Barker K, Boote C, Glaspole I, Goh NSL, Southcott AM, Burge AT, Gillies R, Martin A, Holland AE. The evidence of benefits of exercise training in interstitial lung disease: a randomised controlled trial. Thorax. 2017 Jul;72(7):610-619. doi: 10.1136/thoraxjnl-2016-208638. Epub 2017 Feb 17. PMID 28213592
- [Background] Dowman L, Hill CJ, Holland AE. Pulmonary rehabilitation for interstitial lung disease. Cochrane Database Syst Rev. 2014 Oct 6;(10):CD006322. doi: 10.1002/14651858.CD006322.pub3. PMID 25284270